CLINICAL TRIAL: NCT02649894
Title: Pivotal Multi Center, Randomized, Controlled, Single-Blinded Study Comparing the Silver Nitrate Coated Indwelling Pleural Catheter to the Uncoated PleurX Catheter for the Management of Symptomatic, Recurrent, Malignant Pleural Effusions
Brief Title: Safety and Effectiveness of a New Pleural Catheter for Symptomatic, Recurrent, MPEs Versus Approved Pleural Catheter
Acronym: SWIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS-IP-VH-14-009
Record Dates: First submitted 2015-12-18; First posted 2016-01-08 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Malignant Pleural Effusion
Keywords: malignant pleural effusion
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) (Experimental): Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC)
  Interventions: Device: Experimental: Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC)
- Approved Uncoated PleurX Indwelling Pleural Catheter (Active Comparator): Approved Uncoated PleurX Indwelling Pleural Catheter
  Interventions: Device: Active Comparator: Approved Uncoated PleurX Indwelling Pleural Catheter

INTERVENTIONS:
Device: Active Comparator: Approved Uncoated PleurX Indwelling Pleural Catheter
  Arms: Approved Uncoated PleurX Indwelling Pleural Catheter
Device: Experimental: Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC)
  Other Names: SNCIPC
  Arms: Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC)

SUMMARY:
The purpose of this study is to determine whether a new catheter is safe and effective in treating malignant pleural effusions compared to approve catheter.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, at least 18 years of age, inclusive. 2. Subject has a symptomatic MPE requiring intervention. For an effusion to be defined as malignant, at least one of the following must be true:

  1. There is histocytological confirmation of pleural malignancy
  2. The effusion is an exudate (per Light's criteria) in the context of histocytologically proven malignancy elsewhere, with no other clear cause for fluid identified.

     3. Subject has a history of at least 1 ipsilateral pleural effusion causing dyspnea that responded to thoracentesis where the lung expanded and the dyspnea was improved.

     4. Subject is willing and able to provide written informed consent. 5. Subject is willing and able to meet all study requirements, including follow-up visits and receiving study-related telephone calls.

     6. Subject has sufficient pleural fluid to allow safe insertion of an IPC. 7. Subject has negative pregnancy test if appropriate. 8. Subject or caregiver is able to perform home drainage of the pleural effusion (a caregiver can be a friend, family member or paid healthcare professional and applies to US sites only; UK subjects will have drainage managed by home-care nurses).

     Exclusion Criteria:
* 1. Subject has significant trapped lung, or a proximal bronchial obstruction which is likely to lead to trapped lung. For a subject to be eligible for this study, 2 separate study center clinicians must agree that there is no significant trapped lung on the same CXR using visual estimation (reference guide). The CXR used to make this decision must have been performed ≤30 days preceding the consent form being signed, and must have been performed preferably on the same day, but no more than 7 calendar days after a pleural drainage.

Significant trapped lung is deemed present if any 1 of the following criteria is met:

1. A CXR shows hydropneumothorax.
2. A CXR shows ≥20% of the affected hemithorax to be free of the expected lung parenchymal markings and there is no suggestion of pleural fluid.
3. A CXR shows ≥20% of the affected hemithorax to be occupied with pleural fluid AFTER a pleural aspiration which resulted in symptoms suggestive of trapped lung (e.g., chest pain or cough).

   2. Subject has a Karnofsky score <50, or a World Health Organization (WHO)/ Eastern Cooperative Oncology Group (ECOG) performance status ≥3. Subjects who have a performance status of 3 may be considered for the study if the removal of their fluid would likely improve their performance score by 1 or more.

   3. Subject is pregnant, planning to become pregnant, or is lactating. 4. Subject has a history of empyema. 5. Subject has a history of chylothorax. 6. Subject has an uncorrected coagulopathy. 7. Subject has a hypersensitivity to new or existing pleural catheter or it's components.

   8. Subject has evidence, in the opinion of the Investigator, of either on-going systemic or pleural infection.

   9. Subject has had a lobectomy or pneumonectomy on the side of the effusion. 10. Subject has undergone a previous attempt at ipsilateral pleurodesis which has failed.

   11. Subject has previously been diagnosed with a serious immunodeficiency disorder.

   12. Subject has bilateral pleural effusions, with both being at least moderate in size (greater than one-third of the hemithorax on CXR).

   13. Subject has evidence of fluid loculation such that attempts at pleurodesis are likely to be futile.

   14. Subject has a mediastinal shift of ≥2 cm toward the side of the effusion. 15. Subject is receiving concurrent intrapleural chemotherapy or radiation therapy to the ipsilateral chest.

   16. Subject has any clinical condition, diagnosis, or social circumstance that, in the opinion of the Investigator, would mean participation in the study would be contraindicated.

   17. Subject has no access to a telephone. 18. Subject has no documented blood values (complete blood count [CBC], coagulation tests, urea and electrolytes, and liver function tests [LFTs]) within the last 10 days.

   19. Subject has previously participated in any clinical trial with the investigational device.

   20. Subject currently enrolled in any other clinical investigation or who has participated in any clinical investigation in the 30 days prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-05; Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Shrager, MD, Principal Investigator — Stanford University
Locations (19):
- United States (16):
  - Heart Center Research, Huntsville, Alabama
  - Stanford University School of Medicine/ Stanford Cancer Institute, Stanford, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern Unversity, Chicago, Illinois
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deconess Medical Center West, Boston, Massachusetts
  - Washington Universtiy School of Medicine, Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - SUNY Upstate Hospital, Syracuse, New York
  - UNC Hospital, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Vanderbuilt University, Nashville, Tennessee
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- United Kingdom (3):
  - Southmead Hospital, Bristol
  - Oxford Center for Respiratory Medicine, Churchill Hospital, Oxford
  - Great Western Hospital, Swindon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shrager JB, Bhatnagar R, Kearney CT, Retzlaff NP, Cohen E, Stanton AE, Keyes C, Wahidi MM, Gillespie C, Rahman N, Kerry AL, Feller-Kopman D, Nader D, Akulian J, Chen A, Berry M, Majid A, Reddy C, Tremblay A, Maskell NA. Silver Nitrate-coated versus Standard Indwelling Pleural Catheter for Malignant Effusions: The SWIFT Randomized Trial. Ann Am Thorac Soc. 2022 Oct;19(10):1722-1729. doi: 10.1513/AnnalsATS.202111-1301OC. PMID 35363591

RESULTS

PARTICIPANT FLOW:
Groups:
- Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC): Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC)
  Experimental: Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC)
- Approved Uncoated PleurX Indwelling Pleural Catheter: Approved Uncoated PleurX Indwelling Pleural Catheter
  Active Comparator: Approved Uncoated PleurX Indwelling Pleural Catheter
Period: Overall Study
Arm/Group | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) | Approved Uncoated PleurX Indwelling Pleural Catheter
Started | 81 | 38
Device Inserted | 77 | 37
Completed Day 30 | 56 | 35
Completed (Day 90) | 37 | 27
Not Completed | 44 | 11
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 30 | 7
Not completed — Other, not specified | 6 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) | Approved Uncoated PleurX Indwelling Pleural Catheter | Total
Number analyzed (Participants) | 81 | 38 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.95) | 66.7 (10.35) | 65.4 (10.75)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 35 | 15 | 50
  Gender: Female | 45 | 23 | 68
  Gender: Missing | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 66 | 34 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 64 | 29 | 93
  United Kingdom | 17 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Achieving Pleurodesis Without Recurrence.
Time Frame: 30 days post catheter insertion
Population: All participants who successfully had the catheter placed.
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) | Approved Uncoated PleurX Indwelling Pleural Catheter
Number analyzed (Participants) | 77 | 37
Participants | 17 | 12

2. Secondary Outcome: Time to Confirmed Pleurodesis
Time Frame: 30 days post insertion
Population: Participants who had catheter successfully inserted
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) | Approved Uncoated PleurX Indwelling Pleural Catheter
Number analyzed (Participants) | 77 | 37
days | 11.4 (14.44) | 18.7 (19.3)

3. Secondary Outcome: Time to Recurrence
Description: This endpoint was meant to measure time to recurrence; however, only 1 participant (in the SNCIPC group) had a recurrence so this outcome could not be analyzed.
Time Frame: 90 days post insertion
Population: Participants who had catheter successfully inserted
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) | Approved Uncoated PleurX Indwelling Pleural Catheter
Number analyzed (Participants) | 77 | 37
Participants | 1 | 0

4. Other Pre Specified Outcome: Proportion of Surviving Subjects Without a Trapped Lung Diagnosis Following IPC Placement Who Have Confirmed Pleurodesis Without Recurrence at 14, 30, 60, 90 Days.
Time Frame: Day 14, Day 30, Day 60, Day 90
Population: Participants with catheter successfully placed
Measure: Number; unit: proportion of participants
Arm/Group | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) | Approved Uncoated PleurX Indwelling Pleural Catheter
Number analyzed (Participants) | 77 | 37
proportion of participants
  Day 14 | 0.2222 | 0.2162
  Day 30 | 0.3019 | 0.3333
  Day 60 | 0.3261 | 0.4286
  Day 90 | 0.2500 | 0.5000

5. Other Pre Specified Outcome: Proportion of Subjects With Confirmed Pleurodesis and Without Recurrence 30 Days After IPC Placement by Cancer Type (Lung, Breast and Others).
Time Frame: 30 days.
Population: Participants with successfully placed catheter
Measure: Number; unit: proportion of participants
Arm/Group | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) | Approved Uncoated PleurX Indwelling Pleural Catheter
Number analyzed (Participants) | 77 | 37
proportion of participants
  Lung Cancer | 0.2222 | 0.4545
  Breast Cancer | 0.2000 | 0.1429
  Other Cancer | 0.2273 | 0.3158

6. Other Pre Specified Outcome: Incidence of IPC Occlusion
Time Frame: 90 days
Population: Participants with successfully placed catheter
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) | Approved Uncoated PleurX Indwelling Pleural Catheter
Number analyzed (Participants) | 77 | 37
Participants | 15 | 1

7. Other Pre Specified Outcome: Incidence of Empyema and Cellulitis
Time Frame: 90 days
Population: Participants with successfully placed catheter
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) | Approved Uncoated PleurX Indwelling Pleural Catheter
Number analyzed (Participants) | 77 | 37
Participants | 3 | 2

8. Other Pre Specified Outcome: Pain Using 100 mm Visual Analog Scale (VAS)
Description: Chest pain was measured using a 100 mm VAS scale at baseline and at each subsequent visit. The resulting VAS score ranges from 0 to 100, with 0 indicating "No pain" and 100 indicating "Very severe pain". Therefore, the lower the number, the less chest pain the subject is feeling at the time.
Time Frame: Baseline,Day 7, 14, 30, 45, 75, and 90
Population: Participants with successfully placed catheter
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) | Approved Uncoated PleurX Indwelling Pleural Catheter
Number analyzed (Participants) | 77 | 37
units on a scale
  Baseline | 22.7 (26.63) | 18.0 (26.74)
  Day 7 | 16.9 (26.78) | 10.3 (20.46)
  Day 14 | 9.8 (16.62) | 4.6 (7.82)
  Day 30 | 10.0 (18.53) | 10.2 (19.72)
  Day 45 | 8.4 (17.84) | 8.6 (19.68)
  Day 60 | 10.7 (22.74) | 12.9 (26.48)
  Day 75 | 7.4 (19.97) | 6.4 (17.30)
  Day 90 | 9.6 (18.41) | 9.2 (23.21)

ADVERSE EVENTS:
Time Frame: 90 Days
Description: Participants were monitored for Adverse Events at each study visit (15, 30, 45, 60, 75, 90 days)
Arm/Group | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) | Approved Uncoated PleurX Indwelling Pleural Catheter
All-Cause Mortality (participants affected / at risk) | 30/77 | 7/37
Serious Adverse Events (participants affected / at risk) | 56/77 | 20/37
Other Adverse Events (participants affected / at risk) | 48/77 | 25/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) (N=77) | Approved Uncoated PleurX Indwelling Pleural Catheter (N=37)
Pneumonia (Infections and infestations) | 9 (9) | 3 (4)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Pleural Infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2)
Catheter site infection (Infections and infestations) | 2 (2) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Device breakage (General disorders) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Cerebrovascuar accident (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silver Nitrate Coated Indwelling Pleural Catheter (SNCIPC) (N=77) | Approved Uncoated PleurX Indwelling Pleural Catheter (N=37)
Anaemia (Blood and lymphatic system disorders) | 9 (13) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Catheter site pain (General disorders) | 8 (9) | 4 (4)
Pyrexia (General disorders) | 7 (7) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
C-reactive protein increased (Investigations) | 3 (3) | 2 (2)
Breath sounds abnormal (Investigations) | 1 (1) | 2 (2)
Blood chloride decreased (Investigations) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Large number of deviations (e.g. missed procedures) affected interpretability of data & device performance. Independent adjudication of complex endpoints may have facilitated interpretation, had it been included in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT02649894/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT02649894/SAP_001.pdf